CLINICAL TRIAL: NCT04720053
Title: A Feasibility Study Evaluating Mindfulness-Based Intervention Assessing- A Wearable Wellness Brain Sensing Device (Muse-S) in Newly Diagnosed Fibromyalgia Patients.
Brief Title: Evaluating Mindfulness-Based Interventions With New Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sanjeev Nanda, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-003020
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Wearable brain sensing wellness device headband system (Experimental): Subject diagnosed with fibromyalgia at Mayo Clinic GIM Fibromyalgia Clinic will receive a wearable brain sensing wellness device headband system, and will be given a demonstration of the mindfulness sessions, with detailed instructions on how to begin each session.
  Interventions: Device: Wearable brain sensing wellness device headband system

INTERVENTIONS:
Device: Wearable brain sensing wellness device headband system — Brain sensing headband that measures brain activity by detecting electrical impulses created by the brain.

SUMMARY:
The purpose of this study is to study the feasibility of a wearable brain sensing wellness device to provide mindfulness training to fibromyalgia patients who have failed medical therapy.

DETAILED DESCRIPTION:
All study participants will receive a wearable brain sensing wellness device, and demonstration of the mindfulness sessions. Participants will be asked to complete study surveys/questionnaires. During the first part of study, participants will be asked to complete the intervention. After completion of the intervention they will enter a follow-Up Phase, where they will be contacted and asked to complete surveys and gauge satisfaction with the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent.
* Diagnosed with Fibromyalgia.
* Not pregnant by subject self-report at time of consent.
* Have the ability to provide informed consent.
* Have the ability to complete all aspects of this trial.
* Have access to a iPhone, iPad, Android device.
* Has no contraindicating comorbid health condition as determined by the clinical investigators.

Exclusion Criteria:

* Used or been enrolled in any treatments for fibromyalgia, or pain within the past 30 days.
* Used an investigational drug within the past 30 days.
* Currently (within the past 3 weeks) been practicing mindfulness training on a weekly/regular basis.
* Currently (within the past 3 weeks) been undergoing an additional program (e.g. CAM) to improve quality of life.
* Currently (within 3 weeks) been enrolled in another clinical or research program (e.g. CAM) which intervenes on the patients' QOL, or stress.
* An unstable medical or mental health condition as determined by the physician investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Nanda, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were patients diagnosed with fibromyalgia at a large healthcare facility in the Midwestern United States. Enrollment took place from November 01, 2021 to January 27, 2023. Study participation concluded on July 28, 2023.
Pre-assignment Details: After consent, one participant was found not to meet study entry criteria (no mobile device) and had to be removed from study.
Period: Overall Study
Arm/Group | Wearable Brain Sensing Wellness Device Headband System
Started | 40
Completed | 28
Not Completed | 12
Not completed — Lost to Follow-up | 12

BASELINE CHARACTERISTICS:
Arm/Group | Wearable Brain Sensing Wellness Device Headband System
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  male | 6
  female | 33
  other | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Widespread Pain Index (WPI)
Description: Wide pain index (WPI) defined as a 4-quadrant plus axial pain, measuring widespread pain in 19 body areas where the patient feels pain over the prior week. Each area identified on the list counts as 1. The range on the WPI score can range from 0 to 19. With lower number indicating fewer areas of pain (hence lower pain). The difference is calculated by taking the baseline score minus the end of treatment score.
Time Frame: Baseline to end of treatment (day 90)
Population: Those with complete data at both baseline and end of treatment (day 90)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wearable Brain Sensing Wellness Device Headband System
Number analyzed (Participants) | 28
units on a scale | 1.4 (2.8)

2. Primary Outcome: Change in Perceived Stress Scale
Description: Measured on a 0-10 pain assessment scale. Participants rate their stress on a scale of 0 to 10. Zero means "no stress," and 10 means "the worst possible stress". The difference is calculated by taking the baseline score minus the end of treatment score.
Time Frame: Baseline to end of treatment (day 90)
Population: Participants with measurements at both baseline and end of treatment (day 90)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wearable Brain Sensing Wellness Device Headband System
Number analyzed (Participants) | 30
units on a scale | 4.1 (6.04)

ADVERSE EVENTS:
Time Frame: The time frame was from the start of the study till the end of study, which was a 6 month period.
Description: Adverse Events were collected at the baseline visit and all other visits during the study period. At the end of study visit (6 months) only serious adverse events were collected.
Arm/Group | Wearable Brain Sensing Wellness Device Headband System
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04720053/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/53/NCT04720053/SAP_003.pdf